CLINICAL TRIAL: NCT03754400
Title: A Randomized Controlled Trial of Efficacy of Albumin Therapy With Standard Medical Treatment (SMT) as Compared to Standard Medical Treatment (SMT) in Improving Patient Survival and Immune Modulation in Patients With Acute on Chronic Liver Failure (ASIA Trial).
Brief Title: Efficacy of Albumin Therapy With Standard Medical Treatment (SMT) as Compared to Standard Medical Treatment (SMT) in Improving Patient Survival and Immune Modulation in Patients With Acute on Chronic Liver Failure (ASIA Trial).
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-ACLF-02
Record Dates: First submitted 2018-11-17; First posted 2018-11-27 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Acute on Chronic Liver Failure
MeSH Terms: conditions — Acute-On-Chronic Liver Failure | interventions — Albumins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Albumin (Experimental): All patients will receive a daily intravenous infusion of 20% Human Albumin Solution (HAS) 40 gram at day 0 (loading dose), Day-1 to day 7, 20 gm daily, then from day 8 to day 28, 20 gm every alternate day.
  Interventions: Biological: Albumin; Other: Standard Medical Treatment
- Standard Medical Treatment (Active Comparator): Antibiotics, nutrition and supportive treatment.
  Interventions: Other: Standard Medical Treatment

INTERVENTIONS:
Biological: Albumin — All patients will receive a daily intravenous infusion of 20% Human Albumin Solution (HAS) 40 gram at day 0 (loading dose), Day-1 to day 7, 20 gm daily, then from day 8 to day 28, 20 gm every alternate day.
  Arms: Albumin
Other: Standard Medical Treatment — Antibiotics, nutrition and supportive treatment

SUMMARY:
The AIM of the study is to study the efficacy of intravenous albumin and standard medical treatment as compared to standard medical treatment alone in ameliorating/preventing SIRS and improving survival at 28 days .The project will be conducted in ILBS from august 2018 to December 2019Concept is to understand the immunology, pathophysiology and effects of albumin in the management of ACLF for betterment of the patient's condition and early recovery.

All ACLF patients will be included as per the inclusion and exclusion criteria , after taking informed consent from the patient or their relatives. Will be evaluated for the possible risk factors for the development of SIRS/sepsis in ACLF patients and possible beneficial factors for resolution of SIRS /sepsis in ACLF patients. The effects of albumin administration as per this protocol versus standard medical treatment alone will be reviewed If patient develops allergic reactions to albumin, fluid overload, albumin will be stopped and patient will be treated accordingly to medical condition.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years to 65 years
2. ACLF patients

Exclusion Criteria:

1. Patients who have already received albumin in last 1 week
2. Patients who require albumin like PICD (Paracentesis-Induced Circulatory Dysfunction)

   ,SBP (Spontaneous bacterial peritonitis),LVP(large volume paracentesis),HRS(hepatorenal syndrome)
3. Not given consent
4. Significant cardiopulmonary or structural heart disease/ CKD(chronic kidney diseses) /volume overload /upper GI bleed.
5. Pregnant/ HIV / HCC >2cm size
6. Alcoholic hepatitis eligible for steroids
7. Previous known allergic/adverse reaction to albumin
8. Any clinical condition which the investigator considers would make the patient unsuitable for the trial
9. Patients who will receive palliative treatment only during their hospital admission

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-09-10 (Actual); Primary Completion 2020-07-30 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
Transplant free survival in both groups | 28 days

SECONDARY OUTCOMES:
Transplant free survival in both groups. | 7 days
Incidence or resolution of infection in both groups | 7 day
Incidence or resolution of infection in both groups | 14 day
Incidence or resolution of infection in both groups | 28 day
Number of participant with development of new organ failure in both groups. | 7 day
Number of participant with development of new organ failure in both groups. | 14 day
Number of participant with development of new organ failure in both groups. | 28 day
Adverse events in both groups. | 28 day

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided